CLINICAL TRIAL: NCT03105518
Title: Predictors of Postoperative Pain Following Oocyte Retrieval for Assisted Reproduction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lawrence Ching Tsen, Vice Chair, Faculty Development and Education; Associate Professor, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-P-002310/1
Record Dates: First submitted 2014-10-05; First posted 2017-04-10 (Actual); Results first posted 2017-12-05 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Oocyte Retrieval; Postoperative Pain
Keywords: assisted reproduction; postoperative pain; opioid
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl; Acetaminophen; Oxycodone; oxycodone-acetaminophen

STUDY DESIGN:
Intervention Model Description: Assessment of immediate and delayed postoperative pain
Oversight: Data Monitoring Committee: No

ARMS (1):
- Analgesia options (Experimental): Protocolized analgesia based on VAS degree of discomfort and time. Analgesic options include heating pad, acetaminophen, percocet (oxycodone), fentanyl 0.5-1 mcg/kg.
  Interventions: Drug: Fentanyl; Drug: Acetaminophen; Drug: Oxycodone

INTERVENTIONS:
Drug: Fentanyl — 0.5, 1 mcg/kg
  Other Names: Sublimaze
Drug: Acetaminophen — Single + Oxycodone
  Other Names: Tylenol
Drug: Oxycodone — With Acetaminophen
  Other Names: Percocet

SUMMARY:
The central objective of this study will be to evaluate the relationship between estrogen levels and the pain following oocyte retrieval in women undergoing in vitro fertilization.

DETAILED DESCRIPTION:
Subject will undergo standard clinical protocols for the entire oocyte stimulation cycle and all assisted reproductive procedure decisions and algorithms will be decided entirely independent of this study.

The anesthetic and postoperative pain regimens will use the same agents and dose ranges used in clinical standard practice; however, the regimens will be standardized, so as to limit confounding variables. The study regimen for anesthesia will differ from the current, clinical standard by the mandated use of actual body weight (in current practice, actual, adjusted ideal, or ideal body weights are used), the use of fentanyl 1 mcg/kg IV (instead of 100 mcg for everyone), and the standardization of postoperative analgesia (noted below). The total amount of fentanyl, propofol, and postoperative drugs will be recorded.

Postoperative analgesia will be standardized based on the subject's self reported verbal analogue score (VAS) and the timing of the report. The agents and timing used below differ from the current clinical standard by assessing VAS and responding with a certain regimen.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I to III health status (moderate systemic disease),
* Age between 18 and 50 yrs
* Undergoing oocyte retrieval with intravenous general anesthesia.

Exclusion Criteria:

* Refuse or withdraw their consent
* Fail to adequately respond to IVF stimulations medications, and thus are not eligible for oocyte retrieval.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence C Tsen, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Harnett MJ, Bhavani-Shankar K, Datta S, Tsen LC. In vitro fertilization-induced alterations in coagulation and fibrinolysis as measured by thromboelastography. Anesth Analg. 2002 Oct;95(4):1063-6, table of contents. doi: 10.1097/00000539-200210000-00050. PMID 12351295
- [Result] Bader AM, Datta S, Moller RA, Covino BG. Acute progesterone treatment has no effect on bupivacaine-induced conduction blockade in the isolated rabbit vagus nerve. Anesth Analg. 1990 Nov;71(5):545-8. doi: 10.1213/00000539-199011000-00016. PMID 2221417
- [Result] Datta S, Lambert DH, Gregus J, Gissen AJ, Covino BG. Differential sensitivities of mammalian nerve fibers during pregnancy. Anesth Analg. 1983 Dec;62(12):1070-2. PMID 6650889

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Analgesia Options
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Analgesia Options
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.54 (4.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 95
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 90
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Amount of Discomfort
Description: Change in discomfort following oocyte retrieval with standardized anesthesia management as measured by verbal analogue scoring (0-10 scale). VAS scores correlate to minimal (VAS 0-3), moderate (VAS 4-6) or severe (VAS ≥7) discomfort.
Time Frame: PACU admission, 15, 30 and 60 min postprocedure, postoperative day 3
Population: On PACU admission, subjects were divided into three groups based on the intensity of discomfort. A standardized postoperative analgesic regimen followed, based on VAS score and time (≤ or > than 30 min).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Analgesia Options
Number analyzed (Participants) | 100
units on a scale
  Time 0; ≤10 Follicles: number analyzed (Participants) | 54
  Time 0; ≤10 Follicles | 1.53 (2.13)
  Time 0; > 10 Follicles: number analyzed (Participants) | 46
  Time 0; > 10 Follicles | 3.25 (2.9)
  Time 15; ≤10 Follicles: number analyzed (Participants) | 54
  Time 15; ≤10 Follicles | 2.68 (2.19)
  Time 15; >10 Follicles: number analyzed (Participants) | 46
  Time 15; >10 Follicles | 3.61 (1.98)
  Time 30; ≤10 Follicles: number analyzed (Participants) | 54
  Time 30; ≤10 Follicles | 1.66 (1.40)
  Time 30; >10 Follicles: number analyzed (Participants) | 46
  Time 30; >10 Follicles | 2.93 (1.43)
  Time 60; ≤10 Follicles: number analyzed (Participants) | 54
  Time 60; ≤10 Follicles | 0.97 (1.16)
  Time 60; >10 Follicles: number analyzed (Participants) | 46
  Time 60; >10 Follicles | 2.19 (1.55)
  Time POD 3; ≤ 10 Follicles: number analyzed (Participants) | 54
  Time POD 3; ≤ 10 Follicles | 1.44 (1.15)
  Time POD 3; > 10 Follicles: number analyzed (Participants) | 46
  Time POD 3; > 10 Follicles | 1.64 (1.82)
Statistical Analysis 1: Comparison: Analgesia Options; VAS at Time 0; Follicles ≤10 vs. > 10; Test type: Superiority; p = 0.007, Kruskal-Wallis; 1 way test, chisquare approximation = 7.1880
Statistical Analysis 2: Comparison: Analgesia Options; VAS at Time 15; Follicles ≤10 vs. > 10; Test type: Superiority; p = 0.056, Kruskal-Wallis; 1 way Test, ChiSquare Approximation = 3.6396
Statistical Analysis 3: Comparison: Analgesia Options; VAS at Time 30; Follicles ≤10 vs. > 10; Test type: Superiority; p < 0.0001, Kruskal-Wallis; 1 way Test, ChiSquare Approximation = 15.971
Statistical Analysis 4: Comparison: Analgesia Options; VAS at Time 60; Follicles ≤10 vs. > 10; Test type: Superiority; p < 0.0001, Kruskal-Wallis; 1-way Test, ChiSquare Approximation = 16.0972

2. Secondary Outcome: Amount of Discomfort Following Discharge Until Embryo Transfer
Description: Change in discomfort following oocyte retrieval with standardized anesthesia management as measured by verbal analogue scoring (0-10 scale) after immediate postoperative period (1 hrs) but prior to Embryo Transfer on 3rd postoperative day. Visual Analogue Scale (VAS) scores correlate to minimal (VAS 0-3), moderate (VAS 4-6) or severe (VAS ≥7) discomfort. Patients will record the type, dose, and timing of pain medicines in a diary to be returned at Embryo Transfer.
Time Frame: After 1 hrs but less than 3 days
Population: All 100 parturients analyzed; divided into those who had less than, compared to more than 10 follicles on preoperative ultrasound image.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Analgesia Options
Number analyzed (Participants) | 100
units on a scale
  POD1; ≤10 Folli: number analyzed (Participants) | 54
  POD1; ≤10 Folli | 2.15 (1.72)
  POD1; >10 Follicles: number analyzed (Participants) | 46
  POD1; >10 Follicles | 3.21 (1.87)
  POD2; ≤10 Folli: number analyzed (Participants) | 54
  POD2; ≤10 Folli | 1.28 (1.89)
  POD2; >10 Folli: number analyzed (Participants) | 46
  POD2; >10 Folli | 2.50 (2.35)
Statistical Analysis 1: Comparison: Analgesia Options; VAS at Post Operative Day 1; Follicles ≤10 vs. > 10; Test type: Superiority; p = 0.0991, Kruskal-Wallis; 1-way Test, ChiSquare Approximation = 2.7205
Statistical Analysis 2: Comparison: Analgesia Options; VAS at Post Operative Day 2; Follicles ≤10 vs. > 10; Test type: Superiority; p = 0.2109, Kruskal-Wallis; 1 way Test, ChiSquare Approximation = 1.5654
Statistical Analysis 3: Comparison: Analgesia Options; VAS at Post Operative Day 3; Follicles ≤10 vs. > 10; Test type: Superiority; p = 0.9287, Kruskal-Wallis; 1-way Test, ChiSquare Approximation = 0.0080

ADVERSE EVENTS:
Time Frame: 3 days
Groups:
- Analgesia Options: Protocolized analgesia based on VAS degree of discomfort and time. Analgesic options include heating pad, acetaminophen, percocet (oxycodone), fentanyl 0.5-1 mcg/kg.
  Fentanyl: 0.5, 1 mcg/kg
  Acetaminophen: Single + Oxycodone
  Oxycodone: With Acetaminophen
  No Adverse Events in any subject
Arm/Group | Analgesia Options
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

LIMITATIONS AND CAVEATS:
No limitations or caveats noted for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-09-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT03105518/Prot_SAP_000.pdf